CLINICAL TRIAL: NCT05670366
Title: Proof-of-concept Study for the Integration of Physical Activity Into the Clinical Decision Process of Physically Active People with Type 1 Diabetes
Brief Title: The Integration of Physical Activity Into the Clinical Decision Process of People with Type 1 Diabetes
Acronym: ENHANCED1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: prof dr Pieter Gillard (Other)
Collaborators: University Colleges Leuven Limburg (Unknown)
Responsible Party: Sponsor-Investigator, prof dr Pieter Gillard, Principal investigator, Universitaire Ziekenhuizen KU Leuven
Organization: Universitaire Ziekenhuizen KU Leuven (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: S64550
Record Dates: First submitted 2022-08-29; First posted 2023-01-04 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2024-03

CONDITIONS: Type 1 Diabetes
Keywords: Physical activity; Artificial intelligence
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity | interventions — Fitness Trackers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Physically active participants (Other): There is only one study arm, namely all participants are subjected to the same interventions.
  Interventions: Device: Activity tracker and chest strap; Device: Diary app

INTERVENTIONS:
Device: Activity tracker and chest strap — During the study, the participants will be asked to wear a commercially-available activity tracker during day and night, and a chest strap during sport activities to collect data on physical activity (type, intensity and duration of activity).
Device: Diary app — During the study, the participants will be asked to log the ingestion of carbohydrates, periods and type of physical activity, feelings (e.g. sick, stress, ...) in a diary app.

SUMMARY:
Every person with type 1 diabetes needs personalized advice to integrate physical activity into daily diabetes management. The purpose of this study is to collect data on food intake, physical activity, glucose levels and insulin delivery from people with type 1 diabetes who are physically active. At least 25 people with type 1 diabetes will be asked to perform 25 sports activities of at least half an hour, wear an activity tracker (day and night) and chest strap (during sports activities), and log data on food intake, periods and type of physical activity, and feelings (e.g., sick, stress) in a diary app. Diabetes data such as insulin administration and sensor data will be collected through diabetes management platforms. The primary endpoint involves a database containing data on glucose, insulin administration, physical activity, and food intake of people with type 1 diabetes for statistical analyses and visualizations regarding the relationship between physical activity and blood glucose response.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* 18-80 years old
* Type 1 diabetes ≥1 year
* Using a CGM for more than 6 months
* Using insulin (insulin pens, insulin pumps or hybrid closed-loop systems) to manage glycaemia for more than 6 months
* No use of adjunctive therapies, such as SGLT2-inhibitors or GLP-1 analogues
* No known diabetic gastroparesis
* HbA1c of the last two diabetes consultations are both <10%
* Being physically active at least twice a week on two separate days for 30 consecutive minutes

Exclusion Criteria:

* Age <18 years or >80 years
* People with type 2 diabetes, people with secondary diabetes
* Begin treatment with insulin (insulin pens, insulin pumps or hybrid closed-loop systems) less than 6 months before inclusion
* Not using CGM prior to inclusion
* Known diabetic gastroparesis
* HbA1c > 10% during one of the last two diabetes consultations
* Not willing to use an activity tracker, the diary app or the food app
* Not being physically active on a regular basis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Database which contains insulin data (insulin dose over time) retrieved from diabetes management platforms. | Through study completion (after 25 sport activities), an average of 6 weeks
Database which contains glucose data (glycemic values over time) retrieved from diabetes management platforms. | Through study completion (after 25 sport activities), an average of 6 weeks
Database which contains physical activity data (type of activity) retrieved from the activity tracker and chest strap. | Through study completion (after 25 sport activities), an average of 6 weeks
Database which contains physical activity data (intensity of activity) retrieved from the activity tracker and chest strap. | Through study completion (after 25 sport activities), an average of 6 weeks
Database which contains physical activity data (duration of activity) retrieved from the activity tracker and chest strap. | Through study completion (after 25 sport activities), an average of 6 weeks
Database which contains food intake data (timing of food) retrieved from the diary app. | Through study completion (after 25 sport activities), an average of 6 weeks
Database which contains food intake data (amount of food in grams) retrieved from the diary app. | Through study completion (after 25 sport activities), an average of 6 weeks
Database which contains food intake data (type of food) retrieved from the diary app. | Through study completion (after 25 sport activities), an average of 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Gillard, MD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided